CLINICAL TRIAL: NCT06151613
Title: Non-invasive Electrophysiological Monitoring in High Risk Pregnancies at the Obstetric High Care: the NIEM-O Study
Brief Title: Continuous Non-invasive Electrophysiological Monitoring in High Risk Pregnancies
Acronym: NIEM-O
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxima Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Nadine de Klerk, MD, researcher, PhD candidate, Maxima Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL82869.015.22
Record Dates: First submitted 2023-11-01; First posted 2023-11-30 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Perinatal Outcomes; Preterm Birth; High Risk Pregnancy
Keywords: Electrophysiological monitoring; Cardiotocography; Antepartum monitoring; continuous monitoring; Non-invasive fetal monitoring
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: A single center prospective cohort intervention study with historical controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous eCTG monitoring (Active Comparator): For the continuous eCTG monitoring, a wireless abdominal electrode patch (measuring fetal heart rate (FHR) and uterine activity (UA)) is used, developed by Nemo Healthcare: The Nemo Fetal Monitoring System (NFMS).
  The advantage of the NFMS is that is a safe method for continuous (24/7) fetal monitoring. Furthermore, the patch does not have to be repetitively repositioned during registration, it can be used under the shower and it is wireless giving women more freedom to move around freely. Another benefit of eCTG monitoring is that it is especially suited for women with obesity, where conventional CTG monitoring often fails
  Interventions: Device: continuous eCTG monitoring using the NFMS
- Conventional intermittent CTG monitoring (No Intervention): Conventional intermittent CTG monitoring is performed in Maxima Medical Centre by the use of Philips Avalon FM 30 (Philips Healthcare, Eindhoven, The Netherlands).
  This is a combined external measurement method using two transducers placed on the maternal abdomen: one to measure fetal heart rate (FHR) by the use of Doppler ultrasound (DU) and the other at the fundus of the uterus to measure uterine activity (UA) pattern (TOCO), keeping them in place with elastic banding.

INTERVENTIONS:
Device: continuous eCTG monitoring using the NFMS — Eligible women will be prospectively included in the cohort receiving standard treatment: CTG monitoring intermittent up to three times a day. From these eligible women, a random sample (464) of the prospective cohort (511) will be offered to receive a new monitoring method: 24/7 eCTG monitoring with NFMS. In order to strengthen the comparison between the two groups (eCTG and standard treatment), additional data from 1400 women who received standard treatment in 2014-2019 will be collected retrospectively.
  Arms: Continuous eCTG monitoring

SUMMARY:
The goal of this single centre cohort intervention study with historical controls, is to investigate the effect of implementing continuous antepartum electrophysiological CTG (eCTG) monitoring at the Obstetric High Care (OHC), on perinatal and maternal outcomes and obstetric care.

The main aim is to investigate the effect of both monitoring methods on:

* primary outcome: perinatal outcomes (a composite of perinatal mortality or major neonatal morbidity) until hospital discharge
* secondary outcomes: Maternal mortality, neonatal morbidity, satisfaction for both patient and caregiver, duration of pregnancy, switch of monitoring method, duration of admission to the OHC, timing (planned or emergency) and number of obstetric interventions (such as caesarean section), and admission and duration of admission to the NICU (neonatal intensive care unit).

Eligible women will be prospectively included in the cohort receiving standard treatment: CTG monitoring intermittent up to three times a day. From these eligible women, a random sample (464) of the prospective cohort (511) will be offered to receive a new monitoring method: 24/7 eCTG monitoring. In order to strengthen the comparison between the two groups (eCTG and standard treatment), additional data from 1400 women who received standard treatment in 2014-2019 will be collected retrospectively.

DETAILED DESCRIPTION:
Pregnant women in need for maternal and/or fetal monitoring are hospitalized at the obstetric high care (OHC) of Máxima Medical Center (MMC). They are monitored for up to three times a day with conventional cardiotocography (CTG). In the meantime they reside at the OHC, but the status of the fetus and uterine activity (UA) is not monitored. Nemo Healthcare developed a wireless abdominal electrode patch for measuring fetal heart rate (FHR) and UA: The Nemo Fetal Monitoring System (NFMS). Previous research on non-invasive electrophysiological CTG (eCTG) has yielded promising results in monitoring FHR and UA both during pregnancy and labor. With the use of eCTG technology, safe continuous 24/7 monitoring is possible, which is not possible with conventional cardiotocography. The investigators hypothesize that by introducing continuous antepartum eCTG monitoring perinatal and maternal outcomes will improve.

The investigators aim to include 1911 pregnant women ≥18 years old with a singleton pregnancy between 23+0 and 32+0 weeks of gestation requiring hospitalization on the OHC for maternal or fetal surveillance (including 1400 historical controls).

Additional objectives: The collected NFMS and demographic data will be used to develop and verify a mathematical model for the prediction of time until (preterm) birth, which may be used in clinical practice to reduce unnecessary OHC admissions and facilitate a better timing of interventions. Furthermore, data collected in this study (NFMS, accelerometric, annotated ultrasound) will be used for the development and verification of a mathematical model for the automated detection of fetal movements in NFMS data. This latter model might provide new opportunities in non-invasive monitoring of fetal health.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Singleton pregnancy ≥23+0 weeks of gestation
* Requiring hospitalization to the OHC for maternal or fetal surveillance (i.e. imminent preterm delivery(PPI), PE, HELLP, pregnancy induced hypertension (PIH), FGR, fetal distress, vaginal blood loss, fetal congenital anomalies)
* Parents wishing for fetal monitoring

Exclusion Criteria:

* Multiple pregnancy
* Insufficient knowledge of Dutch or English language
* Contraindications to abdominal patch placement (dermatologic diseases of the abdomen precluding preparation of the abdomen with abrasive paper)
* Women connected to an external or implanted electrical stimulator (e.g. a pacemaker - exclusion due to possible signal interference)
* Fetal and/or maternal cardiac disease (i.e. arrhythmia, congenital defect)
* Treatment plan (with intervention planned within 24 hours after admission) already made before inclusion is completed
* Women admitted with a clinical diagnosis of sepsis with hypotension (i.e. septic shock).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1911 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of perinatal mortality and major neonatal morbidity | during admission (immediately after birth until hospital discharge) or until at least 4 weeks after birth
  A composite outcome consisting of: 1. Incidence of perinatal mortality and/or 2.Incidence of a major neonatal morbidity (defined as either: Intraventricular hemorrhage (IVH) grade three or more, Periventricular leukomalacia (PVL) grade two or more, Moderate or severe bronchopulmonary dysplasia (BPD), Necrotizing enterocolitis (NEC) grade two or more, or Retinopathy of prematurity (ROP) necessitating laser therapy).

SECONDARY OUTCOMES:
Incidence of maternal mortality | From moment of inclusion until six weeks after giving birth
  Incidence of maternal mortality in percentages
Incidence of neonatal morbidity | From inclusion assessed up to 6 months after inclusion
  Incidence of other neonatal morbidity then described in the primary outcome (i.e. IVH grade 1-2, PVL grade 1, mild BPD, NEC grade 1, ROP not necessitating laser therapy, hypoxic ischemic encephalopathy, neonatal seizures, neonatal sepsis (culture proven), need for intubation on the delivery room, mechanical ventilation within the first 72 hours after birth, antibiotics within the first 72 hours after birth, spontaneous intestinal perforation (SIP) necessitating surgery, surfactant treatment, Apgar score <7 after 5 minutes, severe metabolic acidosis (pH <7.05 and base deficit ≥12mmol/L).
Assesment using a surveys (D-QUEST) to measure patient satisfaction | At discharge, assessed up to 1 month.
  Patient satisfaction of the given monitoring method, measured using a surveys: D-QUEST (comprises twelve items with a 5-point rating system. A high level of satisfaction is correlated with a high D-QUEST score, (Score between 14 and 70). The questionnaire is given ones to the patient during the trial.
Assesment using a survey (EQ5D5L) to measure patient satisfaction | EQ5D5L questionnaire is given on day 1 of the admission (day 1 after inclusion). and assessed up to 1 month.
  Patient satisfaction of the given monitoring method, measured using a survey: EQ5D5L (This assessment tool assigns a numerical value to each response level (i.e., 1 for "no problems", 5 for "extreme problems"/"unable to") and the summing of these values across the five items, results in a score. The score is then placed on a scale, which is numbered from 0 to 100. 100 means the best health one can imagine. 0 means the worst health one can imagine). The questionnaire is given ones to the patient during the trial.
Assesment using one survey (Browns survey) to measure caregiver satisfaction | Caregivers are invited to fill in the questionnaire at baseline and at 1 year
  Caregiver satisfaction is measured using Browns survey: purpose of this survey is to assess obstetricians' and midwives' use of current fetal-monitoring techniques and their views towards continuous monitoring, using multiple choice options (ranging from strongly agree to strongly disagree).
Duration of pregnancy in days | Measured from first day of pregnancy until birth, pregnancy period must be related to pregnancy at time of inclusion in the study. Assessed up to 5,5 months after inclusion.
  Duration of pregnancy measured in days
Switch of monitoring method from eCTG to CTG monitoring | From inclusion assessed up to 6 months after inclusion
  Percentage of participants in which a switch is made from eCTG to CTG monitoring
Duration of admission to the Obstetric High Care in days | From inclusion assessed up to 6 months after inclusion
  Duration of admission to the Obstetric High Care measured in days
Timing of obstetric interventions (caesarean section) | From inclusion assessed up to 6 months after inclusion
  Planned or emergency caesarean section
Number of obstetric interventions (caesarean section) | From inclusion assessed up to 6 months after inclusion
  Number of obstetric intervention is measured as number of caesarean sections
Admission (yes/no) to the NICU (neonatal intensive care unit) | From inclusion assessed up to 6 months after inclusion
  Admission to NICU is qualified as yes or no
Duration of admission to the NICU (neonatal intensive care unit) in days. | From inclusion assessed up to 6 months after inclusion
  Duration of admission to the NICU (neonatal intensive care unit) is measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: SG Oei, Prof.dr., Principal Investigator — Maxima Medical Center
Locations (1):
- Maxima Medical Centre, Veldhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Start when IPD is requested
Access Criteria: Anonymous data will be shared to those requesting data published open access, meeting data sharing regulations.

REFERENCES:
- [Derived] de Klerk ND, Berben PBQ, de Vries IR, Niemarkt H, Vullings R, van den Heuvel ER, van der Ven M, Fransen AF, Oei SG, van Laar JOEH. Continuous non-invasive electrophysiological monitoring in high-risk pregnancies: study protocol of a cohort intervention random sampling study in a tertiary obstetrical care centre in the Netherlands (NIEM-O study). BMJ Open. 2025 Nov 12;15(11):e102732. doi: 10.1136/bmjopen-2025-102732. PMID 41224309